CLINICAL TRIAL: NCT07042750
Title: Eccentric Cycling Exercise During Pulmonary Rehabilitation in Patients With Cardiopulmonary Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Silvia Ulrich Somaini (Other)
Collaborators: Klinik Barmelweid (Other)
Responsible Party: Sponsor-Investigator, Silvia Ulrich Somaini, Prof. Silvia Ulrich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EccRehab2
Record Dates: First submitted 2025-06-10; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Eccentric Exercise Training
Keywords: Eccentric cycling exercise; Pulmonary rehabilitation

STUDY DESIGN:
Intervention Model Description: Intervention: Eccentric cycling (instead of usual cycling) + standard care Control: Standard care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric cycling (Experimental): Patients perform eccentric cycling exercise instead of normal cycling exercise in addition to standard car during a cardiopulmonary rehabilitation
  Interventions: Other: Eccentric cycling exercise
- Standard care (Active Comparator): Patients perform cardiopulmonary rehabilitation according to standard care
  Interventions: Other: Standard Care Arm

INTERVENTIONS:
Other: Eccentric cycling exercise — Patients perform eccentric cycling exercise instead of normal cycling exercise in addition to standard car during a cardiopulmonary rehabilitation
  Arms: Eccentric cycling
Other: Standard Care Arm — Patients perform cardiopulmonary rehabilitation according to standard care
  Arms: Standard care

SUMMARY:
Eccentric cycling exercise (ECC) allows training at low metabolic costs and may therefore be valuable for patients with pulmonary vascular disease (PVD). For these patients, regular exercise training has an evidence level 1A recommendation in the current guidelines. Exercise training during longer and regular periods provides chronic adaptation, for which ECC was recently found to have a greater effectiveness than CON by increasing muscle strength, hypertrophy, six-minute walking distance and furthermore, by increasing maximum oxygen uptake (V'O2max) especially in patients with chronic obstructive pulmonary disease (COPD), chronic left heart failure or coronary heart disease. Furthermore, we conducted an RCT in which we exposed patients with PVD to ECC and concluded that ECC is a feasible and well-tolerated exercise modality for PVD patients with severely lower O2 demand and load to the right ventricle. The study in patients with PVD was started (EccRehab), and the great potential was recognized. Therefore there was an indication to open the inclusion criteria to all cardiopulmonary patients with indication for pulmonary rehabilitation (EccRehab2).

For this purpose, the aim of this project is to investigate whether ECC improves exercise capacity and possibly hemodynamics during prolonged rehabilitation programs in patients with cardiopulmonary diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PVD, either PAH or CTEPH via right heart catheterization, according to recent guidelines [9]
* Diagnosed with a cardiopulmonary disease as indication for a pulmonary rehabilitation
* Stable medication for at least 1 month
* Age 18years to 85 years
* No resting hypoxemia (PaO2 >7.3 kPa)
* Medical indication to prescibe a pulmonary rehabilitation

Exclusion Criteria:

* Any co-morbidity that limits the patient to participate the full rehabilitation
* Enrollments in other trials with active treatments
* Language barriers that limits the patient to participate in the rehabilitation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Peak exercise performance [Watts] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  Peak exercise performance is measured during cardiopulmonary exercise tests on a cycle ergometer. The Unit of the measurement is watts.

SECONDARY OUTCOMES:
Peak oxygen uptake [L/min] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  Peak oxygen uptake is measured during cardiopulmonary exercise tests on a cycle ergometer. The Unit of the measurement is liters per minute.
Ventilatory equivalents for carbon dioxide (Minute ventilation / carbon dioxide output) | At baseline pre-intervention and immediately after three weeks of rehabilitation
  Ventilatory equivalents for carbon dioxide is measured during cardiopulmonary exercise tests on a cycle ergometer. The measurement is a ratio without a unit (VE/VCO2).
Six minute walk distance [meters] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The maximal distance that a patient is able to walk within six minutes. The unit of the measurement is meters.
Knee extension test [repetitions] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The patients has to stad up from a chair and sit down as often the patient is able to do this within 1 minute. The unit of the measurement is repetitions.
Systolic pulmonary arterial pressure [mmHg] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The sytolic pulmonary arterial pressure is measured by echocardiography using continuous wave doppler at the tricuspid valve. The unit of the measurement is mmHg.
Total pulmonary reistance [Wood units] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The total pulmonary resistance is measured by echocardiography by dividing the systolic pulmonary arterial pressure by the cardiac output. The unit of the measurement is woos units.
Right ventricular to arterial coupling [mm/mmHg] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The right ventricular arterial coupling is measured by echocardiography dividing the tricuspid annular plane systolic excursion by the systolic arterial pressure. the unit is mm/mmHg.
Cardiac output [L/min] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The cardiac output is measured by echocardiography using the left ventricular outflow tract velocity time integral assessed by pulse wave doppler. The unit of the measurement is L/min.
Arterial partial pressure for oxygen [kPa] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The arterial partial pressure for oxygen is measured by taking a arterial blood sample from the arteria radialis at peak exercise and analyze it in a radiometer. The unit of the measurement is kPa.
Arterial partial pressure for carbon dioxide [kPa] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The arterial partial pressure for carbon dioxide is measured by taking a arterial blood sample from the arteria radialis at peak exercise and analyze it in a radiometer. The unit of the measurement is kPa.
Arterial oxygen saturation [%] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The arterial oxygen saturation is measured by taking a arterial blood sample from the arteria radialis at peak exercise and analyze it in a radiometer. The unit of the measurement is %.
Patient reported leg fatigue [scale from 1 to 10] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  Patients perceived leg fatigue is assessed at peak exercise on the Borg CR 10 scale. The unit of the measurement is a scale from 1 to 10.
Patient reported dyspnea [scale from 1 to 10] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  Patients perceived dyspnea is assessed at peak exercise on the Borg CR 10 scale. The unit of the measurement is a scale from 1 to 10.
Patient reported quality of life [cm] | At baseline pre-intervention and immediately after three weeks of rehabilitation
  The patient reported quality of life is assessed by the visual analogue scale, where the patient has to draw on a 10 cm long line where left is "bad" and right is "very good". The unit of the measurement is cm.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Klinik Barmelweid, Barmelweid
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided